CLINICAL TRIAL: NCT01856517
Title: Up Regulation of Alpha-1 Receptors Upon Septic Shock ?
Brief Title: Upregulation of Alpha-1 Receptors Upon Septic Shock?
Acronym: CATACHOC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Principal Investigator, Eric Dardare, MD attending physician, Direction Centrale du Service de Santé des Armées
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2011PPRC01TURC
Record Dates: First submitted 2013-04-19; First posted 2013-05-17 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Septic Shock
Keywords: pressor response; chronotropic response
MeSH Terms: conditions — Shock, Septic | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): saline administration over 24 h following full optimization of patient according to current guidelines
  Interventions: Drug: Placebo
- clonidine (Active Comparator): clonidine 1 mcg.kg-1.h-1 over 24 h following full optimization of the patient according to current guidelines
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine
  Arms: clonidine
Drug: Placebo
  Arms: placebo

SUMMARY:
The hallmarks of septic shock are hypovolemia and reduced pressor response to endogenous noradrenaline. The working hypothesis is that the higher the plasma concentration of endogenous noradrenaline will be, the lower the pressor response to exogenous noradrenaline will be. This will be tested in patients presenting with septic shock, following state of the art management (including repeated assessment of vena cava diameter and compliance, and response to dynamic indices of loading) following placebo vs clonidine administration (1 mcg.kg-1.h-1 over 24 h without bolus) and administration of increasing doses of noradrenaline (1 mcg, 2 mcg, etc. up to a delta systolic blood pressure circa 25-30 mm Hg).

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to the CCU with septic shock : SBP<90 mm Hg refractory to volume load (>30 ml.kg-1 within 6 h before inclusion) thus in need administration of noradrenaline for >1 h (0.1 mcg.kg-1.h-1 i.e. >0.5 mg.h-1/70 kg) to maintain mean BP>65 mm Hg.
* criteria for sepsis :temperature>38.5 or <36°C ; WBC>12 000 or <4000/ml ; tachypnea (>20 cycles par min) or mechanical ventilation ; tachycardia : >90 bpmin
* written informed consent by the patient or next of kin or signature by the investigators of the form "emergency inclusion"

Exclusion Criteria:

* age<18 ans
* pregnancy
* mental illness making informed consent impossible
* Absence of consent as signed by the patient or next of kin or signature of "emergency inclusion form"
* individual without social security coverage or participating in another biomedical research
* Contre-indications to clonidine (uncorrected hypovolemia, sick sinus syndrom, III grade AV block)
* HR<70 bp/min
* pre-exitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
change in pressor response to exogenous noradrenaline | 0 and 24 h
  bolus of exogenous noradrenaline (1 mcg and up) are administered to the patient to evoke an increase in delta systolic blood pressure by 25-30 mm Hg. Administration of increasing dose of noradrenaline is stopped as soon as delta systolic blood pressure has reached 25-30 mm Hg.

SECONDARY OUTCOMES:
change in heart rate response to increasing doses of dobutamine (100 mcg and up) to evoke an increase in heart rate up to 20 beats per min. | 0 and 24 h

CONTACTS AND LOCATIONS:
Locations (1):
- Critical Care Unit, Hopital Desgenettes, Lyon, France